CLINICAL TRIAL: NCT00537628
Title: Biomarkers in Acute Heart Failure: An International, Multi-Center Trial Evaluating the Prognostic and Diagnostic Utility of Biomarkers in Patients With Heart Failure Presenting With Shortness of Breath
Brief Title: Biomarkers in Acute Heart Failure
Acronym: BACH
Status: Completed | Type: Observational
Sponsor: Brahms AG (Industry)
Responsible Party: Andreas Bergmann, PhD Chief Research Officer, BRAHMS AG
Other Study IDs: Brahms
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Shortness of Breath; Heart Failure
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objectives

1. Mid Region pro Adrenomedullin (MR-proADM) is superior to BNP for the prognosis of heart failure (HF) patients and adds incremental value in predicting outcomes for patients presenting to the Emergency Department (ED) with shortness of breath.
2. Mid Region pro A-Type Natriuretic Peptide (MR-proANP) is non-inferior to BNP for the diagnosis of HF in patients presenting to the ED with shortness of breath.

DETAILED DESCRIPTION:
The diagnosis of heart failure is often very difficult. Clinical history is often vague, and physical examination findings suffer from lack of specificity and sensitivity. For example, symptoms like shortness of breath and edema are often present in patients without cardiac disease, while elevated jugular venous pressure can be difficult to visualize and auscultation of a third heart sound can be challenging to hear, especially in an emergency room setting.

Although BNP levels can sometimes help clarify the clinical picture when patients present acutely with shortness of breath, patients both with and without heart failure may have BNP values that fall into a "gray zone", where the diagnosis is still very much in question. Also, there can be difficulties in interpreting BNP levels in patients with renal dysfunction, patients with a high body mass index, and patients of advanced age.

Investigative tests in the emergency department such as the electrocardiogram or chest x-ray are also non-specific for diagnosing heart failure. Tests such as echocardiography, while accurate in the assessment of left ventricular dysfunction, are expensive and are not always available on an emergent basis; furthermore, the presence of heart failure with normal systolic function (a.k.a. diastolic dysfunction) can complicate the interpretation of echocardiograms. Additionally, just because a patient has systolic dysfunction on an urgent echocardiogram does not mean that their acute dyspnea is due to heart failure, and so the test itself may not accurately reflect the acute situation at hand.

Another difficult diagnostic dilemma arises when a patient with a history of heart failure presents with signs that could also be consistent an acute respiratory illness such as pneumonia. Often, patients with background heart failure have elevated BNP levels at baseline. In this setting, chest radiographs can be especially difficult to interpret when one must distinguish between edema and infiltrates, or possibly both.

For all of these reasons, there is a pressing need for additional tools to help us differentiate heart failure from other causes of dyspnea in our acutely short of breath patients, and to improve our ability to provide accurate prognostic information and sound therapeutic management to our heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older.
* The patients must be seen in the urgent care or emergency area with a chief complaint of shortness of breath not due to trauma.

Exclusion Criteria:

* Patient is unable to sign or understand the consent form.
* Patient is on any dialysis.
* Patient has trauma related shortness of breath (i.e. penetrating wounds, crush injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 1641 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Maisel, MD, Principal Investigator — Veterans Affairs Medical Center, San Diego and University of California, San Diego; Stefan D Anker, MD, PhD, Principal Investigator — Universitätsklinikum Charité, Charité - Campus Virchow; Frank Peacock, MD, Study Chair — The Cleveland Clinic
Locations (15):
- United States (8):
  - University of California, San Diego, San Diego, California
  - Veterans Affairs Medical Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Cleveland Clinic, Cleveland, Ohio
  - Virgina Commonwealth University, Richmond, Virginia
- Charite- Universitatsmedizin Berlin, Berlin, Germany
- Athens University Hospital Attikon, Athens, Greece
- University La Sapienza, Rome, Italy
- University of Otago, Christchurch, New Zealand
- Clinical Military Hospital, Wroclaw, Poland
- University Hospital Basel, Basel, Switzerland
- University of Leicester, Leicester, United Kingdom

REFERENCES:
- [Derived] Maisel A, Neath SX, Landsberg J, Mueller C, Nowak RM, Peacock WF, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Clopton P, Filippatos GS, Di Somma S, Anand I, Ng LL, Daniels LB, Christenson RH, Potocki M, McCord J, Terracciano G, Hartmann O, Bergmann A, Morgenthaler NG, Anker SD. Use of procalcitonin for the diagnosis of pneumonia in patients presenting with a chief complaint of dyspnoea: results from the BACH (Biomarkers in Acute Heart Failure) trial. Eur J Heart Fail. 2012 Mar;14(3):278-86. doi: 10.1093/eurjhf/hfr177. Epub 2012 Feb 2. PMID 22302662
- [Derived] Peacock WF, Nowak R, Christenson R, DiSomma S, Neath SX, Hartmann O, Mueller C, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Filippatos GS, Anand I, Ng LL, Daniels LB, Morgenthaler N, Anker SD, Maisel AS. Short-term mortality risk in emergency department acute heart failure. Acad Emerg Med. 2011 Sep;18(9):947-58. doi: 10.1111/j.1553-2712.2011.01150.x. PMID 21906204
- [Derived] Maisel A, Mueller C, Nowak RM, Peacock WF, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Clopton P, Filippatos GS, Di Somma S, Anand I, Ng LL, Daniels LB, Neath SX, Christenson R, Potocki M, McCord J, Hartmann O, Morgenthaler NG, Anker SD. Midregion prohormone adrenomedullin and prognosis in patients presenting with acute dyspnea: results from the BACH (Biomarkers in Acute Heart Failure) trial. J Am Coll Cardiol. 2011 Aug 30;58(10):1057-67. doi: 10.1016/j.jacc.2011.06.006. PMID 21867843
- [Derived] Maisel A, Xue Y, Shah K, Mueller C, Nowak R, Peacock WF, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Clopton P, Filippatos GS, Di Somma S, Anand IS, Ng L, Daniels LB, Neath SX, Christenson R, Potocki M, McCord J, Terracciano G, Kremastinos D, Hartmann O, von Haehling S, Bergmann A, Morgenthaler NG, Anker SD. Increased 90-day mortality in patients with acute heart failure with elevated copeptin: secondary results from the Biomarkers in Acute Heart Failure (BACH) study. Circ Heart Fail. 2011 Sep;4(5):613-20. doi: 10.1161/CIRCHEARTFAILURE.110.960096. Epub 2011 Jul 15. PMID 21765124
- [Derived] Maisel A, Mueller C, Nowak R, Peacock WF, Landsberg JW, Ponikowski P, Mockel M, Hogan C, Wu AH, Richards M, Clopton P, Filippatos GS, Di Somma S, Anand I, Ng L, Daniels LB, Neath SX, Christenson R, Potocki M, McCord J, Terracciano G, Kremastinos D, Hartmann O, von Haehling S, Bergmann A, Morgenthaler NG, Anker SD. Mid-region pro-hormone markers for diagnosis and prognosis in acute dyspnea: results from the BACH (Biomarkers in Acute Heart Failure) trial. J Am Coll Cardiol. 2010 May 11;55(19):2062-76. doi: 10.1016/j.jacc.2010.02.025. PMID 20447528